CLINICAL TRIAL: NCT06937710
Title: Analysis of Biomechanical Parameters and Return to Sport After Hip Arthroscopy
Acronym: ATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Sport, Bordeaux Mérignac (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-62-SBM
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hip Arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomechanical analysis (Experimental)
  Interventions: Diagnostic Test: Measure of symmetry between the inferior limbs

INTERVENTIONS:
Diagnostic Test: Measure of symmetry between the inferior limbs — Hip force moments will be analyzed in the 3 planes (in Nm/Kg) and compared between the two legs.

SUMMARY:
The aim of this prospective study is to describe dynamic movement parameters in active patients who underwent surgery between 3 and 6 months after hip arthroscopy, focusing on movements such as jumping, squatting and acceleration. By examining the relationships between these different parameters and the return to sporting activities, and by integrating different angle and alignment measurements per- and post-operatively, we hope to find predictive factors for successive rehabilitation in athletes, which could lead to more personalized rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Hip arthroscopy for labrum lesion
* athlete prior to arthroscopy with desire to return to sport

Exclusion Criteria:

* Previous surgery or pathology of the operated lower limb
* Contralateral hip operated
* Neurological pathology affecting movement
* Medical condition contraindicating participation in sports
* Dementia or inability to complete questionnaires and assessments
* Pregnant or breast-feeding patient
* Patient under protective supervision
* Patient not covered by a social security scheme

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Symmetry of hip muscular forces between the two lower limbs | 3 months after surgery ; 6 months after surgery
  Hip force moments will be measured in 3 planes (sagittal, frontal, transverse), in Nm/Kg, using a set of sensors and force and pressure platforms.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport Bordeaux Merignac, Mérignac, France

IPD SHARING:
Plan to Share IPD: No